CLINICAL TRIAL: NCT06635161
Title: Neuromodulation With Transcranial Pulse Stimulation of the Anterior Insula Cortex and Dorsal Anterior Cingulate Cortex in Healthy Adults: A Randomized, Single-blind, Three-arm, Sham-controlled, Pilot Trial
Brief Title: Trancranial Pulse Stimulation on Anterior Insula Cortex and Dorsal Anterior Cingulate Cortex
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Principal Investigator, Dr Georg Kranz, Principal Investigator, The Hong Kong Polytechnic University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HSEARS20240319006
Record Dates: First submitted 2024-10-02; First posted 2024-10-10 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2025-06

CONDITIONS: Healthy Adults

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- TPS on AIC (Experimental): 1. Healthy adults aged 18-65 years old will receive ten sessions of real TPS (1000 pulses per session) on the bilateral anterior insula cortex (AIC) within 2 weeks (5 sessions per week). 2. Before and after TPS, participants will perform four psychological tasks (the reading the mind in the eyes test, the balloon analog risk task, the Go/No-go task, the counting stroop task). 3. The stimulation target on the bilateral AIC will be determined by transforming MNI coordinates (left AIC: x=-41, y=6, z=3; right AIC: x=44, y=9, z=2) into the individual T1-weighted space. 4. To optimize the penetration depth of TPS pulses, a standard stand-off device (Neurology) will be used when stimulating AIC.
  Interventions: Device: Transcranial pulse stimulation (with Neurology stand-off device)
- TPS on dACC (Experimental): 1. Healthy adults aged 18-65 years old will receive ten sessions of real TPS (1000 pulses per session) on the bilateral dorsal anterior cingulate cortex (dACC) within 2 weeks (5 sessions per week). 2. Before and after TPS, participants will perform four psychological tasks (the reading the mind in the eyes test, the balloon analog risk task, the Go/No-go task, the counting stroop task). 3. The stimulation target on the bilateral dACC will be determined by transforming MNI coordinates (left dACC: x=-4, y=26, z=45; right dACC: x=7, y=30, z=40) into the individual T1-weighted space. 4. To optimize the penetration depth of TPS pulses, no stand-off device will be used when stimulating dACC.
  Interventions: Device: Trancranial pulse stimulation (without a stand-off device)
- sham TPS on vertex (Sham Comparator): 1. Healthy adults aged 18-65 years old will receive ten sessions of sham TPS (1000 pulses per session) on the vertex within 2 weeks (5 sessions per week). 2. Before and after TPS, participants will perform four psychological tasks (the reading the mind in the eyes test, the balloon analog risk task, the Go/No-go task, the counting stroop task). 3. The stimulation target on the vertex will be determined by transforming MNI coordinates (x=0, y=-30, z=60) into the individual T1-weighted space. 4. A sham stand-off device will be used when stimulating the vertex.
  Interventions: Device: Transcranial pulse stimulation (with a sham stand-off device)

INTERVENTIONS:
Device: Trancranial pulse stimulation (without a stand-off device) — A single session of TPS will be performed, applying 1000 pulses in the session (single ultrashort (3 μs) ultrasound pulses, 0.2 mJ mm-2, 4 Hz pulse frequency). No stand-off device will be used to target dorsal anteior cingulate cortex.
  Arms: TPS on dACC
Device: Transcranial pulse stimulation (with Neurology stand-off device) — A single session of TPS will be performed, applying 1000 pulses in the session (single ultrashort (3 μs) ultrasound pulses, 0.2 mJ mm-2, 4 Hz pulse frequency). A Neurology stand-off device will be used to target the anterior insula cortex.
  Arms: TPS on AIC
Device: Transcranial pulse stimulation (with a sham stand-off device) — A single session of TPS will be performed, applying 1000 pulses in the session (single ultrashort (3 μs) ultrasound pulses, 0.2 mJ mm-2, 4 Hz pulse frequency). A sham stand-off device will be used to target vertex.
  Arms: sham TPS on vertex

SUMMARY:
Transcranial pulse stimulation (TPS) is a newly developed non-invasive brain stimulation (NIBS) technique from Austria & Germany with highly promising applicability in neuropsychiatric disorders. Clinical trials have shown a beneficial effect of TPS in patients with Alzheimer's disease and depression. Although TPS has the capability to noninvasively target deeper brain regions such as the dorsal anterior cingulate cortex (dACC) and anterior insula cortex (AIC), no TPS study has been conducted to investigate the feasibility and effectiveness of dACC or AIC stimulation. Here, a randomized, single-blind, sham-controlled clinical pilot trial is proposed to probe the effects of TPS over bilateral dACC and AIC on modulating cognitive, behavioral and emotional functions and functional connectivity of brain circuits.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 65
* Biological and mental health, based on a clinical interview
* Able to understand and follow instructions by the study team

Exclusion Criteria:

* Major internal diseases, neurological disorders, or mental disorders
* Having a metal implant in the brain
* Corticosteroid treatment within 6 weeks prior to inclusion
* Pregnancy or breastfeeding
* Common NIBS and MRI exclusion criteria, such as a history of brain surgery, cardiac pacemaker, deep brain stimulation, and intracranial metallic particles
* Previous TPS experience
* Color blindness

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 66 (Estimated)
Dates: Start 2024-08-05 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
The Chinese version of reading the mind in the eyes test | Baseline, midpoint (2 weeks after the first TPS session), endpoint (4 weeks after the first TPS session)
  The Chinese version of reading the mind in the eyes test (RMET) will be used to assess the AIC function of empathy. In this test, participants will be presented with a series of 28 photographs of the eye region of the face, followed by four mental state terms. Participants will be asked to choose which of four words best describes what the person in the photograph is thinking, feeling, and expressing. The order of trial presentation within each run will be randomized. Participants will be told to complete the task as quickly as possible although they are not timed.
The Balloon Analog Risk Task | Baseline, midpoint (2 weeks after the first TPS session), endpoint (4 weeks after the first TPS session)
  The Balloon Analog Risk Task will be used to assess the AIC function of risky decision-making. Participants have to inflate a virtual balloon that can either grow larger or explode. Each time participants pump up the balloon, they accumulate money, but each pump also carries the risk of the balloon exploding, which results in the participant losing all of their money from that balloon. In the task, participants will be required to complete 30 trials (balloons) with a maximum of 12 pumps. The probability of explosion will be increased with each pump from 2% for the first pump to 90% for the last pump.
The Go/No-go task | Baseline, midpoint (2 weeks after the first TPS session), endpoint (4 weeks after the first TPS session)
  The Go/No-go task (GNGT) will be used to assess the AIC and ACC function of response inhibition. The red circles and blue circles will serve as Go and No-go signals, respectively. Each trial will begin with the central fixation cross for a duration of 1000 ms, followed by a Go or No-go stimulus for 400 ms. A total of 100 trials will be randomly presented in two blocks, including high (50%) and low (20%) No-go trials. The participants will be instructed to respond as quickly as possible to the Go signal by pressing the space key on the keyboard with the right index finger and to withhold the response when a No-go signal appears. Before the test task, there will be a practice session with 20 trials. At the end of each trial in the test task, participants will receive feedback for 1000 ms indicating their answer is correct or not.
The counting Stroop task | Baseline, midpoint (2 weeks after the first TPS session), endpoint (4 weeks after the first TPS session)
  The counting Stroop task conflict will be used to assess the dACC function of the error monitoring. Participants will be required to report, via key-press, the number of identical words they see on a monitor, regardless of the word's meaning, as quickly and accurately as possible. The alphabets (A, S, K, L) on the keyboard correspond to the number of words (A to 1, S to 2, K to 3, L to 4). In incongruent blocks, the stimuli consisted of Chinese number words such as "一", "二", "三" and "四", while the number of words and meaning will be always inconsistent. During the neutral blocks, Chinese words such as "了", "人", "手", "口" which are irrelevant to the number will be displayed. Both sets of stimuli are common Chinese words with matched visual complexity. Each stimulus will change every 1.5 seconds. The inter-trial interval will be 500 ms. The task consisted of four 48-second blocks of 24 neutral trials alternating with four 48-second blocks of 24 incongruent trials.

SECONDARY OUTCOMES:
Magnetic resonance imaging measurement | baseline (one week before the 1st TPS session), endpoint (4 weeks after the first TPS session)
  Participants will receive a 5-minute structural MRI scan using a Siemens 3T MAGNETOM Prisma system and a 64-channel head coil. The standard scanning parameters will be: TR/TE=2300/2.98 ms, flip angle = 9°, FOV=240x256x208 mm, voxel size=1x1x1 mm. A rs-fMRI scan of 8 minutes will be performed, during which subjects will be instructed to relax with eyes open and gaze at a cross displayed on the screen in front of them, allowing their mind to wander without focusing on anything specific. Rs-fMRI will be performed using a single-shot gradient-recalled EPI with TR/TE=607/32 ms, a FOV of 220x220x160 mm, and a voxel size of 2.5x2.5x2.5 mm with 64 slices (slice thickness = 2.5mm, interleaved series).

CONTACTS AND LOCATIONS:
Overall Officials: Georg S Kranz, PhD, Principal Investigator — The Hong Kong Polytechnic University
Locations (1):
- The Hong Kong Polytechnic University, Hong Kong, Hung Hom, Kowloon, Hong Kong

IPD SHARING:
Plan to Share IPD: No